CLINICAL TRIAL: NCT00415714
Title: A Randomized Controlled Pilot Trial Testing the Safety and Efficacy of an Ambulatory Biofeedback Device for Primary Insomnia
Brief Title: Safety and Efficacy of an Ambulatory Biofeedback Device for Primary Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helicor (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H300
Record Dates: First submitted 2006-12-21; First posted 2006-12-25 (Estimated); Last update posted 2007-01-29 (Estimated); Status verified 2006-12

CONDITIONS: Primary Insomnia
Keywords: Primary Insomnia; Chronic Insomnia; Biofeedback; Sleeplessness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

INTERVENTIONS:
Device: Portable Biofeedback

SUMMARY:
The objective of this study is to determine the efficacy of a portable biofeedback device on improving sleep latency and other sleep variables such as nocturnal awake time and daytime functioning in persons with primary insomnia.

DETAILED DESCRIPTION:
There is evidence that when compared to normal controls, persons with insomnia exhibit increased cognitive and physiological arousal and higher overall metabolic rate during sleep, particularly at sleep onset. There is evidence that reducing this arousal may impact sleep latency and nocturnal awake time. Although relaxation treatments have been integrated into behavioral therapies, there are numerous barriers to their implementation in real world settings. The present study is designed to examine the effect of a portable biofeedback device designed to induce physiological relaxation as compared to an inactive sham control device condition in reducing sleep onset latency in persons with primary insomnia over a 4 week period at three separate research sites.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18-55
2. Met DSM-IV-TR criteria for Primary Insomnia as measured by the:

   * Structured Interview for Sleep Disorders.
   * Insomnia Severity Index (>14).
3. Demonstrate Sleep Onset Latency of >=45 minutes on >= 3 nights per week greater than or equal to 6 days over the 2 week period.
4. A mean SOL >= 30 minutes over the 2 week period between Screening and Baseline visits.
5. Residential stability (1 year) and means to travel to appointments.
6. Willing to provide the name and contact information of a secondary contact person.
7. Off insomnia medications for at least one week prior to randomization and no more than 2 days of use during the first week of baseline.
8. Ability to read in English.
9. Provision of informed consent.
10. Willing to comply with daily protocol.
11. Ability to obtain a reading on the device.

Exclusion Criteria:

1. Been in more than 2 studies in the past 2 years
2. Pregnant
3. Terminal, progressive, and or unstable medical illness.
4. Self-reported sleep disruptive medical disorder i. Chronic Pain, Fibromyalgia, Pheochromocytoma, Hyperthyroidism, Congestive Heart Failure, Chronic Obstructive Pulmonary Disease, Diabetes.
5. Current Axis I psychiatric disorder.(DSM-IV) i. Major Depressive Disorder, Depression, Generalized Anxiety Disorder, Attention Deficit Disorder, Post Traumatic Stress Disorder, Bipolar Disorder, Substance/Alcohol Use Disorders, Attention Deficit Hyperactivity Disorder, Schizophrenia/Psychotic Disorders, Delirium, Dementia, and/or Amnesic disorders, Panic Disorder w/ nocturnal panic attacks.
6. Chronic alcohol use not diagnosed in criterion 6. i. Subjects unwilling to limit their alcohol intake to 2 standard drinks per day will be excluded.
7. Raynaud's Disease
8. Regularly taking anti-anxiety medications, beta blockers or other heart medications that regulate heartbeat, bronchodilators, respiratory stimulants, simulating antidepressants, sedating antidepressants, thyroid supplements, anti-psychotics, and/or steroids.
9. Regularly taking antidepressants (Prozac, Zoloft, Paxil) and NOT on a fixed dosage for at least 1 month prior to entering the study.
10. Regularly taking medication (prescribed or over the counter) for sleep difficulties (>3x week). Sleep medications include any substance for sleep not limited to but including FDA approved sleep medications, analgesics, antihistamines, decongestants, melatonin, L-trypotophan, and velarian.
11. Unwilling to abstain from PRN sleep aides (prescribed or over the counter).
12. Restless Leg Syndrome as assessed by structured interview.
13. Symptoms of Sleep Apnea (BMI>32 and Epworth Sleepiness Scale >10)
14. Own a negative air ionizer or have used one in the past to treat insomnia.
15. If subject recognizes device during the ability to obtain a pulse rate wave reading on the device.
16. More than 5 cups (8oz) of caffeinated drinks per day and/or unwilling to limit caffeine in-take to a maximum of 3 cups a day and not after 5pm during the intervention.
17. Regular night-time shift work and rotating night-time shift work.
18. Idiopathic Insomnia.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132
Dates: Start 2006-09; Study Completion 2007-10

PRIMARY OUTCOMES:
Sleep latency at 4 week follow-up

SECONDARY OUTCOMES:
wake time after sleep onset (WASO) at 4 week follow-up
total awake time (SOL + WASO) at 4 week follow-up
Shifting from moderate/severe insomnia to mild/no insomnia (Insomnia Severity Index)at 4 week follow-up
Daytime functioning at 4 week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jack Edinger, Ph.D., Principal Investigator — Duke Unversity Medical Center; Charles Morin, Ph.D., Principal Investigator — University of Laval
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Morin CM, Hauri PJ, Espie CA, Spielman AJ, Buysse DJ, Bootzin RR. Nonpharmacologic treatment of chronic insomnia. An American Academy of Sleep Medicine review. Sleep. 1999 Dec 15;22(8):1134-56. doi: 10.1093/sleep/22.8.1134. PMID 10617176
- See also: Sleep website — http://www.aasmnet.org/